CLINICAL TRIAL: NCT06197451
Title: Validity and Reliability of a Turkish Version of MD Anderson Dysphagia Inventory for Neurogenic Patients
Brief Title: Validity and Reliability of a Turkish Version of MD Anderson Inventory Dysphagia Inventory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Assistant Professor, Gazi University
Other Study IDs: 187765
Record Dates: First submitted 2023-12-17; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Dysphagia; Neurologic Disorder
MeSH Terms: conditions — Deglutition Disorders; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients who are diagnosed with neurologic disorders The first group consists of 170 diagnosed with neurologic disorders who have at least six months of dysphagia complaints. The participants will given the Turkish version of M.D. Anderson Dysphagia Inventory, consisted of 20 questions, Swallowing Quality-of-Life Questionnaire and Mini Mental Questionnaire. After the two weeks, 50 participants will given the MDADI for sampling.
  Interventions: Other: Turkish Version of M. D. Anderson Dysphagia Inventory
- 2: Healthy subjects The second group consists of 50 healty participants will given the MDADI consists of 20 questions and Swallowing Quality-of-Life Questionnaire.
  Interventions: Other: Turkish Version of M. D. Anderson Dysphagia Inventory

INTERVENTIONS:
Other: Turkish Version of M. D. Anderson Dysphagia Inventory — Turkish Validation and Cultural Adaptation of M. D. Anderson Dysphagia Inventory in Neurologic Patients

SUMMARY:
The purpose of this study is to M.D. Validity of the Turkish version of the Anderson Dysphagia Inventory for the Turkish population, reliability, and cultural adaptation.

DETAILED DESCRIPTION:
Oropharyngeal dysphagia (OD) is a common finding in patients with neurogenic disorders.

Swallowing disorder can be acute or chronic in nature. For example, acute OD is observed in patients after stroke, head trauma, neurosurgical intervention, or in patients with Guillain-Barré syndrome. Chronic OD may develop in patients who do not recover after a stroke. Degenerative OD, Parkinson's disease, amyotrophic lateral sclerosis, myasthenia gravis, Huntington's disease, myotonic dystrophy type 1 and multiple sclerosis It is seen in patients with progressive neurological diseases. The prevalence of OD in neurogenic patients varies from 3% to 50% in stroke patients and up to almost 100% in patients with Huntington's disease. The OD can lead to weight loss, malnutrition, social isolation, aspiration pneumonia, and reduced health-related quality of life (QoL). Some studies have reported that dysphagia-specific QoL is weakly associated with OD severity measured using, among other things, fiberoptic endoscopic evaluation of swallowing (FEES) and videofluoroscopy of swallowing (VFS). Therefore, dysphagia-specific QoL questionnaires used alongside these instrumental assessments add value by providing insight into patients' perception of OD, which can be taken into account in the treatment plan. There are dysphagia-specific quality-of-life questionnaires that are actively used today: Swallowing Quality of Life Questionnaire (SWAL-QOL, 44 items), Swallowing Disability Index (30 items), Dysphagia Handicap Index (25 items) and M.D. Anderson Dysphagia Inventory (MDADI, 20 items). Multidisciplinary dysphagia clinics in our country mostly focus on the head and neck. It is visited by patients with OD of oncological or neurological origin.The M. D. Anderson dysphagia inventory is an easier inventory to perform since it has a smaller number of questions and contains more standard questions compared to other currently used questionnaires. Other questionnaires, such as the SWAL-QOL-TR and the Swallowing Disability Index, are longer than the MDADI and take more time to complete. The purpose of this study is M.D. Validity of the Turkish version of the Anderson Dysphagia Inventory for the Turkish population, reliability and cultural adaptation.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Diagnosed with neurologic disorder
* Able to speak, read, understand and write in Turkish
* History of dysphagia during 6 months

Group 2:

* Able to speak, read, understand and write in Turkish
* Healthy adults

Exclusion Criteria:

* Mini Mental State Examination score below 23 points
* History of head and neck cancer (HNC),
* Age below 18 or above 85 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosed with neurologic disorder and having oropharyngeal dysphagia and healthy adults
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-02-19 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
Turkish Version of M. D. Anderson Dysphagia Inventory | Baseline
  The M.D Anderson Dysphagia Inventory is a self-administered, psychometrically validated dysphagia-specific questionnaire for cancer patients that is designed to assess the impact of dysphagia on health-related quality of life . Like the original English version, the validated Turkish translation of the M.D. Anderson Dysphagia Inventory consists of 20 items pooled in 4 subscales: the global scale
  (1 item); the functional scale (5 items); the physical scale (8 items); and the emotional scale (6 items)The global question was scored individually, and the mean score of each subscale (emotional, physical, and functional) was multiplied by 20 to obtain a total score with a range from zero (extremely low functioning) to 100 (high functioning). A higher M. D. Anderson Dysphagia Inventory score is indicative of better day-to-day functioning and quality of life.
Turkish Version of M. D. Anderson Dysphagia Inventory | Two weeks
  The M.D Anderson Dysphagia Inventory is a self-administered, psychometrically validated dysphagia-specific questionnaire for cancer patients that is designed to assess the impact of dysphagia on health-related quality of life . Like the original English version, the validated Turkish translation of the M.D. Anderson Dysphagia Inventory consists of 20 items pooled in 4 subscales: the global scale
  (1 item); the functional scale (5 items); the physical scale (8 items); and the emotional scale (6 items)The global question was scored individually, and the mean score of each subscale (emotional, physical, and functional) was multiplied by 20 to obtain a total score with a range from zero (extremely low functioning) to 100 (high functioning). A higher M. D. Anderson Dysphagia Inventory score is indicative of better day-to-day functioning and quality of life.

SECONDARY OUTCOMES:
The Swallowing Quality-of-Life Questionnaire | Baseline
  The Swallowing Quality-of-Life Questionnaire was designed to evaluate the impact of dysphagia on health-related quality of life in dysphagic patients. It consists of 44 items divided among 11 domains: general burden (2 items); food selection (2 items); eating duration (2 items); eating desire (3 items); fear of eating (4 items); sleep (2 items); fatigue (3 items); communication (2 items); mental health (5 items); social functioning (5 items); and frequency of symptoms (14 items). Each item is scored on a 5-point scale: the higher the score, the better the swallow-related quality of life. Completion of the questionnaire takes 15-30 min. The Turkish version of the Swallowing Quality of Life is considered the gold standard for determining dysphagia specific quality of life in patients with dysphagia.

OTHER OUTCOMES:
Subject Demographics and Medical History | Baseline
  The median values of age and ratio of gender in all groups. Medical Diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation Recruiting Ankara, Turkey, 06500, Ankara, Turkey (Türkiye)